CLINICAL TRIAL: NCT03500952
Title: Family Planning Ahead
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: High incidence of fraudulent enrollment.
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Principal Investigator, Rachel L. Thompson, Assistant Professor, The Dartmouth Institute, Dartmouth-Hitchcock Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 00030871
Record Dates: First submitted 2018-04-10; First posted 2018-04-18 (Actual); Last update posted 2019-01-09 (Actual); Status verified 2019-01

CONDITIONS: Contraception; Pregnancy Related

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patient Decision Aid (Experimental): Birth Control After Pregnancy patient decision aid and supporting document
  Interventions: Other: Birth Control After Pregnancy
- Patient Information Leaflet (Active Comparator): Postpartum Birth Control patient information leaflet
  Interventions: Other: Postpartum Birth Control

INTERVENTIONS:
Other: Birth Control After Pregnancy — A 27-page patient decision aid in portable document format (and an accompanying 3-page supporting document in portable document format) hosted online.
  Arms: Patient Decision Aid
Other: Postpartum Birth Control — A 4-page patient information leaflet in portable document format and text format hosted online.
  Arms: Patient Information Leaflet

SUMMARY:
Family Planning Ahead is a study that aims to improve decision-making about postpartum contraception. Family Planning Ahead will test two different strategies: a patient decision aid and a patient information leaflet.

ELIGIBILITY:
Inclusion Criteria:

* Currently pregnant
* Between 28 and 38 weeks' gestation at the time of enrollment
* Estimated due date in March, April, May, or June 2018
* 15 years or older
* Can read and write English
* Live in the United States
* Share a valid email address for study purposes

Exclusion Criteria

* Not currently pregnant
* Less than 28 weeks' or more than 38 weeks' gestation at the time of enrollment
* Estimated due date earlier than March 2018 or later than June 2018
* Under 15 years
* Can not read and write English
* Do not live in the United States
* Do not share a valid email address for study purposes

Min Age: 15 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2018-03-22 (Actual); Primary Completion 2018-08-23 (Actual); Study Completion 2018-08-23 (Actual)

PRIMARY OUTCOMES:
Perceived support in decision-making | T2 (Approximately 7-11 weeks after self-reported estimated due date)
  The extent to which the person feels they received adequate support and advice without pressure to make a decision about postpartum contraceptive methods, measured using adapted versions of the Support subscale of the Decisional Conflict Scale (O'Connor, 1993).

SECONDARY OUTCOMES:
Perceptions of being informed | T0 (immediately following study enrollment); T1 (one week following study enrollment)
  The extent to which the person feels informed of available postpartum contraceptive methods and the benefits, risks, and side effects of each, measured using an adapted version of the Informed subscale of the Decisional Conflict Scale (O'Connor, 1993).
Values clarity | T0 (immediately following study enrollment); T1 (one week following study enrollment)
  The extent to which the person feels clear about personal values related to postpartum contraceptive method benefits, risks, and side effects, measured using an adapted version of the Values Clarity subscale of the Decisional Conflict Scale (O'Connor, 1993).
Decisional uncertainty | T0 (immediately following study enrollment); T1 (one week following study enrollment)
  The extent to which the person feels certain about which postpartum contraceptive method to choose, measured using an adapted version of the Uncertainty subscale of the Decisional Conflict Scale (O'Connor, 1993).
Decision self-efficacy | T0 (immediately following study enrollment); T1 (one week following study enrollment)
  The extent to which the person has self-confidence or belief in their ability to make decisions about postpartum contraceptive methods, measured using an adapted version of the Decision Self-Efficacy Scale (O'Connor, 1995).
Intended contraceptive method(s): LARC vs. other | T0 (immediately following study enrollment); T1 (one week following study enrollment)
  The proportion of people who intend to use a long-acting reversible contraceptive (LARC) method (i.e., hormonal intrauterine device, copper intrauterine device, or implant) 'in the first few months after giving birth', measured using a self-developed item.
Intended contraceptive method(s): Most or moderately effective vs. other | T0 (immediately following study enrollment); T1 (one week following study enrollment)
  The proportion of people who intend to use a most or moderately effective contraceptive method (i.e., female sterilization, hormonal intrauterine device, copper intrauterine device, implant, injection, combined pill, progestin-only pill, patch, ring, diaphragm) 'in the first few months after giving birth', measured using a self-developed item.
Intended contraceptive method(s): Method vs. no method or unsure | T0 (immediately following study enrollment); T1 (one week following study enrollment)
  The proportion of people who intend to use one or more contraceptive methods (i.e., female sterilization, hormonal intrauterine device, copper intrauterine device, implant, injection, combined pill, progestin-only pill, patch, ring, diaphragm, male condom, internal (female) condom, spermicide, sponge, cervical cap, lactational amenorrhea method, withdrawal, fertility awareness, male sterilization, and/or emergency contraceptive pill) 'in the first few months after giving birth', measured using a self-developed item.
Intended timing of contraceptive method(s) initiation: Not unsure vs. unsure | T0 (immediately following study enrollment); T1 (one week following study enrollment)
  The proportion of people who are not unsure about how soon after giving birth they will (first) start using a contraceptive method (i.e., intend to start using a contraceptive method 'in the first 10 minutes', 'in the first few days', 'in the first few weeks', 'around 6 weeks', 'in the first few months' or 'other'), measured using a self-developed item.
Values concordance of intended contraceptive method(s) | T0 (immediately following study enrollment); T1 (one week following study enrollment)
  The proportion of people who perceive optimal values concordance of their intended postpartum contraceptive method(s) (or intention to use no contraceptive methods), measured using the Measure of Alignment of Choices (Thompson et al., 2017).
Trust in health professional(s) | T2 (Approximately 7-11 weeks after self-reported estimated due date)
  The extent to which the person feels trust in the health professional(s) they talk to about postpartum contraception during and/or after pregnancy, measured using an adapted version of the Patient Trust in a Physician Scale (Dugan et al., 2005).
Interpersonal quality of family planning care | T2 (Approximately 7-11 weeks after self-reported estimated due date)
  The proportion of people who report high interpersonal quality of family planning care during and/or after pregnancy, measured using an adapted version of the four-item Interpersonal Quality of Family Planning Care (IQFP-R) scale (Dehlendorf et al. 2016).
Shared decision-making | T2 (Approximately 7-11 weeks after self-reported estimated due date)
  The extent to which which the person feels they experienced shared decision-making about postpartum contraceptive methods during and/or after pregnancy, measured using the CollaboRATE measure (Barr et al., 2014).
Concordance between preferred and actual decision-making involvement (self): Concordant vs. discordant | T2 (Approximately 7-11 weeks after self-reported estimated due date)
  The proportion of people who report concordance between their actual and preferred involvement in the decision to use their postpartum contraceptive method(s), measured using two self-developed items.
Concordance between preferred and actual decision-making involvement (partner): Concordant vs. discordant | T2 (Approximately 7-11 weeks after self-reported estimated due date)
  The proportion of people who report concordance between the actual involvement of their partner and their preferences pertaining to partner involvement in the decision to use their postpartum contraceptive method(s), measured using two self-developed items.
Concordance between preferred and actual decision-making involvement (health professional(s)): Concordant vs. discordant | T2 (Approximately 7-11 weeks after self-reported estimated due date)
  The proportion of people who report concordance between the actual involvement of their health professional(s) and their preferences pertaining to health professional involvement in the decision to use their postpartum contraceptive method(s), measured using two self-developed items.
Time pressure in decision-making | T2 (Approximately 7-11 weeks after self-reported estimated due date)
  The extent to which the person feels they had (or have) enough time to make a decision about postpartum contraceptive methods, measured using a self-developed item.
Pressure to use a certain contraceptive method | T2 (Approximately 7-11 weeks after self-reported estimated due date)
  The extent to which the person felt (or feels) pushed to use a certain postpartum contraceptive method, measured using a self-developed item.
Values concordance of contraceptive method(s) used | T2 (Approximately 7-11 weeks after self-reported estimated due date)
  The proportion of people who perceive optimal values concordance of the postpartum contraceptive method(s) they have used, measured using the Measure of Alignment of Choices (Thompson et al., 2017).
Effective decision | T2 (Approximately 7-11 weeks after self-reported estimated due date)
  The extent to which the person feels they made an effective decision about postpartum contraceptive methods, measured using an adapted version of the Effective Decision subscale of the Decisional Conflict Scale (O'Connor, 1993).
Contraceptive method(s) prescribed in first 60 days: LARC vs. other | T2 (Approximately 7-11 weeks after self-reported estimated due date)
  The proportion of people who report being given or prescribed a long-acting reversible contraceptive (LARC) method (i.e., hormonal intrauterine device, copper intrauterine device, or implant) in the first 60 days after giving birth, measured using a self-developed item.
Contraceptive method(s) prescribed in first 60 days: Most or moderately effective vs. other | T2 (Approximately 7-11 weeks after self-reported estimated due date)
  The proportion of people who report being given or prescribed a most or moderately effective contraceptive method (i.e., female sterilization, hormonal intrauterine device, copper intrauterine device, implant, injection, combined pill, progestin-only pill, patch, ring, diaphragm) in the first 60 days after giving birth, measured using a self-developed item.
Contraceptive method(s) prescribed in first 3 days: LARC vs. other | T2 (Approximately 7-11 weeks after self-reported estimated due date)
  The proportion of people who report being given or prescribed a long-acting reversible contraceptive (LARC) method (i.e., hormonal intrauterine device, copper intrauterine device, or implant) in the first 3 days after giving birth, measured using a self-developed item.
Contraceptive method(s) prescribed in first 3 days: Most or moderately effective vs. other | T2 (Approximately 7-11 weeks after self-reported estimated due date)
  The proportion of people who report being given or prescribed a most or moderately effective contraceptive method (i.e., female sterilization, hormonal intrauterine device, copper intrauterine device, implant, injection, combined pill, progestin-only pill, patch, ring, diaphragm) in the first 3 days after giving birth, measured using a self-developed item.
Contraceptive method(s) used: LARC vs. other | T2 (Approximately 7-11 weeks after self-reported estimated due date)
  The proportion of people who, at the time of survey completion, report having used a long-acting reversible contraceptive (LARC) method (i.e., hormonal intrauterine device, copper intrauterine device, or implant) since giving birth, measured using a self-developed item.
Contraceptive method(s) used: Most or moderately effective vs. other | T2 (Approximately 7-11 weeks after self-reported estimated due date)
  The proportion of people who, at the time of survey completion, report having used a most or moderately effective contraceptive method (i.e., female sterilization, hormonal intrauterine device, copper intrauterine device, implant, injection, combined pill, progestin-only pill, patch, ring, diaphragm) since giving birth, measured using a self-developed item.
Contraceptive method(s) used: Method vs. no method | T2 (Approximately 7-11 weeks after self-reported estimated due date)
  The proportion of people who, at the time of survey completion, report having used one or more contraceptive methods (i.e., female sterilization, hormonal intrauterine device, copper intrauterine device, implant, injection, combined pill, progestin-only pill, patch, ring, diaphragm, male condom, internal (female) condom, spermicide, sponge, cervical cap, lactational amenorrhea method, withdrawal, fertility awareness, male sterilization, and/or emergency contraceptive pill) since giving birth, measured using a self-developed item.
Timing of decision about contraceptive method(s): During pregnancy vs. since giving birth | T2 (Approximately 7-11 weeks after self-reported estimated due date)
  The proportion of people who report deciding to use their postpartum contraceptive method(s) during pregnancy, measured using a self-developed item.
Likelihood of recommending the intervention to a friend | T1 (one week following study enrollment)
  The proportion of people who report that they are extremely likely to recommend the intervention to a friend, measured using a self-developed item.
Likelihood of reviewing the intervention in the future | T1 (one week following study enrollment)
  The proportion of people who report that they are extremely likely to review the intervention in the future, measured using a self-developed item.
Perceived utility of the intervention | T1 (one week following study enrollment)
  The extent to which the person perceives that the intervention was useful in preparing them to communicate with their health professional and make a decision, measured using an adapted version of the Preparation for Decision Making Scale (Graham & O'Connor, 2010).

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Thompson, PhD, Principal Investigator — Dartmouth College
Locations (1):
- Internet (Dartmouth College), Lebanon, New Hampshire, United States

IPD SHARING:
Plan to Share IPD: Yes
The investigators will make an anonymized copy of the final participant-level data set available to others for research purposes, either via data sharing on request or digital repository deposit.

REFERENCES:
- [Background] Dehlendorf C, Henderson JT, Vittinghoff E, Grumbach K, Levy K, Schmittdiel J, Lee J, Schillinger D, Steinauer J. Association of the quality of interpersonal care during family planning counseling with contraceptive use. Am J Obstet Gynecol. 2016 Jul;215(1):78.e1-9. doi: 10.1016/j.ajog.2016.01.173. Epub 2016 Jan 28. PMID 26827879
- [Background] Thompson R, Manski R, Donnelly KZ, Stevens G, Agusti D, Banach M, Boardman MB, Brady P, Colon Bradt C, Foster T, Johnson DJ, Li Z, Norsigian J, Nothnagle M, Olson AL, Shepherd HL, Stern LF, Tosteson TD, Trevena L, Upadhya KK, Elwyn G. Right For Me: protocol for a cluster randomised trial of two interventions for facilitating shared decision-making about contraceptive methods. BMJ Open. 2017 Oct 22;7(10):e017830. doi: 10.1136/bmjopen-2017-017830. PMID 29061624
- [Background] Dugan E, Trachtenberg F, Hall MA. Development of abbreviated measures to assess patient trust in a physician, a health insurer, and the medical profession. BMC Health Serv Res. 2005 Oct 3;5:64. doi: 10.1186/1472-6963-5-64. PMID 16202125
- [Background] Barr PJ, Thompson R, Walsh T, Grande SW, Ozanne EM, Elwyn G. The psychometric properties of CollaboRATE: a fast and frugal patient-reported measure of the shared decision-making process. J Med Internet Res. 2014 Jan 3;16(1):e2. doi: 10.2196/jmir.3085. PMID 24389354
- [Background] Bennett C, Graham ID, Kristjansson E, Kearing SA, Clay KF, O'Connor AM. Validation of a preparation for decision making scale. Patient Educ Couns. 2010 Jan;78(1):130-3. doi: 10.1016/j.pec.2009.05.012. Epub 2009 Jun 26. PMID 19560303
- [Background] O'Connor, A. M. (1995). Decision Self Efficacy Scale: User manual. Retrieved from https://decisionaid.ohri.ca/docs/develop/User_Manuals/UM_Decision_SelfEfficacy.pdf
- [Background] O'Connor, A. (2010). Decisional Conflict Scale: User manual. Retrieved from https://decisionaid.ohri.ca/docs/develop/User_Manuals/UM_Decisional_Conflict.pdf